CLINICAL TRIAL: NCT00417677
Title: A Phase I/II Study of Temsirolimus and Sunitinib in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A Study Combining Treatment With Temsirolimus and Sunitinib for Subjects With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision was made not to attempt a lower dose
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3066K1-402
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-10

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

INTERVENTIONS:
Drug: Combination of Temsirolimus and Sunitinib

SUMMARY:
This study is being conducted to determine the Maximum Tolerated Dose (MTD) and efficacy of the combined treatment of Temsirolimus and Sunitinib for the treatment of Advanced Kidney Cancer

DETAILED DESCRIPTION:
A study to determine the safety, tolerability, and maximum tolerated dose (MTD) of the combination of temsirolimus and sunitinib in subjects with advanced Renal Cell Carcinoma (RCC) (dose escalation phase). Once the MTD is determined, this study will also evaluate the efficacy of this combination by determining progression free survivial (PFS) at 12 months in subjects with advanced RCC (expanded cohort phase).

ELIGIBILITY:
Inclusion Criteria for Dose Escalation Phase

1. Histologically confirmed advanced RCC.
2. Up to 2 prior systemic regimens for RCC.
3. Subject must have at least 1 measurable lesion that can be accurately measured in at least 1 dimension with the longest diameter ³10 mm when measured by spiral computed CT (5-mm slice thickness contiguous) or ³20 mm when measured by conventional CT (10-mm slice thickness contiguous) (lesion must be ³ 2 times the size of the slice thickness per RECIST).

   * More criteria apply

Exclusion Criteria for Dose Escalation Phase

1. Subjects with known active central nervous system (CNS) malignancy (primary or metastatic).
2. Prior therapy with sirolimus, temsirolimus or sunitinib.
3. Subjects receiving known strong Cytochrome P450 (CYP)3A4 isoenzyme inhibitors and/or inducers. Subjects receiving other CYP3A4 isoenzyme inhibitors and/or inducers not classified as strong inhibitors or inducers are eligible, provided they have been on a stable regimen for at least 4 weeks before screening.

   * More criteria apply

Inclusion Criteria for Expanded Cohort Phase

1. Subjects with histologically confirmed advanced RCC regardless of nephrectomy status who have received no prior systemic therapies for their disease.
2. Subjects with histologically confirmed advanced RCC regardless of nephrectomy status who have a least 4 weeks since prior treatment with palliative radiation therapy, and/or surgery and resolution of all toxic effects of prior therapy to NCI CTCAE (version 3.0) grade £1.
3. Subjects must have at least 1 measurable lesion that can be accurately measured in at least 1 dimension with the longest diameter ³10 mm when measured by spiral CT (5-mm slice thickness contiguous) or ³20 mm when measured by conventional CT (10-mm slice thickness contiguous) (lesion must be ³2 times the size of the slice thickness per RECIST).

   * More Criteria apply

Exclusion Criteria for the Expanded Cohort Phase

1. Subjects with a history of a CNS malignancy or metastatic disease to the CNS and subjects with a known, active CNS malignancy (primary or metastatic).
2. Prior anti-vascular endothelial growth factor (anti-VEGF) therapies (with either monoclonal antibodies and/or tyrosine kinase inhibitors [TKIs]) and/or mTOR inhibitors.
3. Subjects receiving known strong CYP3A4 isoenzyme inhibitors and/or inducers. Subjects taking other CYP3A4 isoenzyme inhibitors and/or inducers not classified as strong inhibitors or inducers are eligible, provided they have been on a stable regimen for at least 4 weeks before screening.

   * More Criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2007-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Initially, an ascending dose design will be used in order to evaluate the tolerability and safety of the combination and to determine the MTD of this combination (dose escalation phase)
Once appropriate doses of each agent have been determined, an expanded cohort of 100 subjects with advanced RCC will be enrolled and treated at the MTD, to obtain further safety and efficacy information

SECONDARY OUTCOMES:
To examine additional efficacy endpoints including: Response rate (RR), Overall Survival (OS), & Progression Free Survival at 6 months and 24 months.
To determine the pharmacokinetic (PK) parameters of temsirolimus alone and temsirolimus and sunitinib in combination
PK samples will be collected from 20 subjects in the expanded cohort. Concentrations of temsirolimus, sirolimus, and sunitinib will be analyzed using a noncompartmental modeling approach.The PK parameters will include estimation of the peak concentr

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (4):
- United States (4):
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Philadelphia, Pennsylvania